CLINICAL TRIAL: NCT04217031
Title: Decision Variability Between Different Heart Teams for Complex Coronary Artery
Brief Title: Decision Variability Between Different Heart Teams for Complex Coronary Artery Diseases
Status: Completed | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2019-1303
Record Dates: First submitted 2019-12-31; First posted 2020-01-03 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Coronary Artery Disease
Keywords: Heart team; Decision making; Complex coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Decision variability assessment group: Patients with angiographically confirmed 3-vessel or left main disease will be enrolled. Patients data and heart team decision will be collected to analyze the variability between different heart team decisions.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The purposes of this study are 1) to explore the variability of decisions between different heart teams in complex coronary artery disease; 2) to evaluate the reasons of the discrepancy in decision making.

DETAILED DESCRIPTION:
Heart team has been recommended by guideline for optimizing the decision making for patients with complex coronary artery diseases (CAD). However, prior studies have demonstrated that heart team decision might have poor reproducibility, and the variability of heart team decision remains unknown.

Thus, the investigators designed a single-center, retrospective, cross-sectional study to explore the decision variability of heart team in CAD patients. The investigators will retrospectively recruit patients with angiographically confirmed 3-vessel or left main disease from a coronary angiography database at Fuwai hospital. Patients' baseline information will be collected. And different heart teams will be established and made decisions for the enrolled patients. First, the investigators will assess the decision variability between different heart teams. Secondary, the investigators will evaluate the reason of discrepancy by qualitative and quantitative analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with angiographically confirmed 3-vessel disease or left main disease

Exclusion Criteria:

* Prior percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG)
* Myocardial infarction with acute phase judged by Electrocardiograph or biomarkers
* Combined with severe valvular disease, great vessel disease or huge ventricular aneurysm which need surgery
* Combined with atrial fibrillation or severe arrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients will be randomly selected and enrolled from a coronary angiography registry database at Fuwai hospital to make sure the representativity of enrolled patients.
Sampling Method: Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Kappa value of decisions | at the end of enrollment (6 months)
  Kappa value of decisions between different heart teams

SECONDARY OUTCOMES:
Concordance rate of decisions | at the end of enrollment (6 months)
  Concordance rate of decisions between different heart teams

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No